CLINICAL TRIAL: NCT05525195
Title: Influence of Preoperative Fibrinogen Levels on Blood Loss and Transfusions in Pediatric Cardiac Surgery
Brief Title: Influence of Preop Fibrinogen on Blood in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of department, anesthesiology, Brugmann University Hospital
Other Study IDs: card_ped_fibri
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cardiac Surgery; Congenital Heart Disease; Cardiopulmonary Bypass; Fibrinogenemia
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Congenital cardiac surgery — All children who underwent congenital cardiac surgery with cardiopulmonary bypass between 2008 and 2018

SUMMARY:
Fibrinogen plays an important role in the coagulation cascade. Low levels of preoperative fibrinogen have been associated in adults with higher blood and transfusion requirements during surgery. Guidelines from the European Society of Anesthesiology and Intensive Care recommends fibrinogen substitution based on viscoelastic tests in adult cardiac surgery. Cardiopulmonary bypass results in a profound hemodilution and dilution of all coagulation factors. This is especially true in children where the priming volume of the cardiopulmonary bypass circuit is much higher compared to the patient's weight than in adults. Cardiopulmonary bypass generates high levels of tissue plasminogen activator resulting in a hyperfibrinolysis, further lowering fibrinogen levels.

The aim of this retrospective study is to explore a possible relationship between preoperative fibrinogen levels and perioperative blood loss, as well as transfusion requirements in children undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* all children with cardiac surgery under cardiopulmonary bypass between 2008 and 2018
* Age < 16 year

Exclusion Criteria:

* preoperative coagulopathy
* Jehovah's witnesses
* patients with fresh frozen plasma in the priming of the cardiopulmonary bypass circuit

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children under 16 year, with cardiac surgery under cardiopulmonary bypass between 2008 and 2018 at our institution
Sampling Method: Non-Probability Sample
Enrollment: 932 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Blood loss | Day 0
  Blood loss in mL during surgery and postoperatively during the first 24h (day 0) will be extracted from our database
Transfusion requirements | Day 0
  Transfusion requirements of packed red cells ( in mL), fresh frozen plasma (in mL) and platelets (in mL) during the first 24h (day 0) will be extracted from our database

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Wenderickx, MSc, Study Director — HUDERF
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weisel JW, Litvinov RI. Fibrin Formation, Structure and Properties. Subcell Biochem. 2017;82:405-456. doi: 10.1007/978-3-319-49674-0_13. PMID 28101869
- [Background] Grottke O, Mallaiah S, Karkouti K, Saner F, Haas T. Fibrinogen Supplementation and Its Indications. Semin Thromb Hemost. 2020 Feb;46(1):38-49. doi: 10.1055/s-0039-1696946. Epub 2019 Oct 1. PMID 31574543
- [Background] Corum LE, Hlady V. The effect of upstream platelet-fibrinogen interactions on downstream adhesion and activation. Biomaterials. 2012 Feb;33(5):1255-60. doi: 10.1016/j.biomaterials.2011.10.074. Epub 2011 Nov 17. PMID 22100981
- [Background] Guzzetta NA, Miller BE. Principles of hemostasis in children: models and maturation. Paediatr Anaesth. 2011 Jan;21(1):3-9. doi: 10.1111/j.1460-9592.2010.03410.x. Epub 2010 Sep 16. PMID 20849450
- [Background] Charbonneau H, Pasquie M, Mayeur N. Preoperative plasma fibrinogen level and transfusion in cardiac surgery: a biphasic correlation. Interact Cardiovasc Thorac Surg. 2020 Nov 1;31(5):622-625. doi: 10.1093/icvts/ivaa153. PMID 33137819
- [Background] Kozek-Langenecker SA, Ahmed AB, Afshari A, Albaladejo P, Aldecoa C, Barauskas G, De Robertis E, Faraoni D, Filipescu DC, Fries D, Haas T, Jacob M, Lance MD, Pitarch JVL, Mallett S, Meier J, Molnar ZL, Rahe-Meyer N, Samama CM, Stensballe J, Van der Linden PJF, Wikkelso AJ, Wouters P, Wyffels P, Zacharowski K. Management of severe perioperative bleeding: guidelines from the European Society of Anaesthesiology: First update 2016. Eur J Anaesthesiol. 2017 Jun;34(6):332-395. doi: 10.1097/EJA.0000000000000630. PMID 28459785
- [Background] Faraoni D, Willems A, Savan V, Demanet H, De Ville A, Van der Linden P. Plasma fibrinogen concentration is correlated with postoperative blood loss in children undergoing cardiac surgery. A retrospective review. Eur J Anaesthesiol. 2014 Jun;31(6):317-26. doi: 10.1097/EJA.0000000000000043. PMID 24503704
- [Background] Paparella D, Brister SJ, Buchanan MR. Coagulation disorders of cardiopulmonary bypass: a review. Intensive Care Med. 2004 Oct;30(10):1873-81. doi: 10.1007/s00134-004-2388-0. Epub 2004 Jul 24. PMID 15278267
- [Background] Ravn HB. Hemostasis in Pediatric Cardiac Surgery. Semin Thromb Hemost. 2017 Oct;43(7):682-690. doi: 10.1055/s-0037-1603365. Epub 2017 Jun 8. No abstract available. PMID 28597463
- [Background] Walden K, Jeppsson A, Nasic S, Backlund E, Karlsson M. Low preoperative fibrinogen plasma concentration is associated with excessive bleeding after cardiac operations. Ann Thorac Surg. 2014 Apr;97(4):1199-206. doi: 10.1016/j.athoracsur.2013.11.064. Epub 2014 Feb 6. PMID 24507940
- [Background] Gielen C, Dekkers O, Stijnen T, Schoones J, Brand A, Klautz R, Eikenboom J. The effects of pre- and postoperative fibrinogen levels on blood loss after cardiac surgery: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2014 Mar;18(3):292-8. doi: 10.1093/icvts/ivt506. Epub 2013 Dec 6. PMID 24316606
- [Background] Ranucci M, Jeppsson A, Baryshnikova E. Pre-operative fibrinogen supplementation in cardiac surgery patients: an evaluation of different trigger values. Acta Anaesthesiol Scand. 2015 Apr;59(4):427-33. doi: 10.1111/aas.12469. Epub 2015 Jan 20. PMID 25600583
- [Background] Ranucci M, Bianchi P, Cotza M, Beccaris C, Silvetti S, Isgro G, Giamberti A, Baryshnikova E. Fibrinogen levels and postoperative chest drain blood loss in low-weight (<10 kg) children undergoing cardiac surgery. Perfusion. 2019 Nov;34(8):629-636. doi: 10.1177/0267659119854246. Epub 2019 Jun 28. PMID 31250738
- [Background] Spiezia L, Di Gregorio G, Campello E, Maggiolo S, Bortolussi G, Stellin G, Simioni P, Vida V. Predictors of postoperative bleeding in children undergoing cardiopulmonary bypass: A preliminary Italian study. Thromb Res. 2017 May;153:85-89. doi: 10.1016/j.thromres.2017.03.021. Epub 2017 Mar 22. PMID 28359027
- [Background] Willems A, Patte P, De Groote F, Van der Linden P. Cyanotic heart disease is an independent predicting factor for fresh frozen plasma and platelet transfusion after cardiac surgery. Transfus Apher Sci. 2019 Jun;58(3):304-309. doi: 10.1016/j.transci.2019.03.014. Epub 2019 Mar 19. PMID 30904398
- [Background] Bhardwaj V, Malhotra P, Hasija S, Chowdury UK, Pangasa N. Coagulopathies in cyanotic cardiac patients: An analysis with three point - of - care testing devices (Thromboelastography, rotational thromboelastometry, and sonoclot analyzer). Ann Card Anaesth. 2017 Apr-Jun;20(2):212-218. doi: 10.4103/aca.ACA_4_17. PMID 28393783
- [Background] Van der Linden P, Dumoulin M, Van Lerberghe C, Torres CS, Willems A, Faraoni D. Efficacy and safety of 6% hydroxyethyl starch 130/0.4 (Voluven) for perioperative volume replacement in children undergoing cardiac surgery: a propensity-matched analysis. Crit Care. 2015 Mar 17;19(1):87. doi: 10.1186/s13054-015-0830-z. PMID 25886765
- [Background] Lacroix J, Hebert PC, Hutchison JS, Hume HA, Tucci M, Ducruet T, Gauvin F, Collet JP, Toledano BJ, Robillard P, Joffe A, Biarent D, Meert K, Peters MJ; TRIPICU Investigators; Canadian Critical Care Trials Group; Pediatric Acute Lung Injury and Sepsis Investigators Network. Transfusion strategies for patients in pediatric intensive care units. N Engl J Med. 2007 Apr 19;356(16):1609-19. doi: 10.1056/NEJMoa066240. PMID 17442904
- [Background] Willems A, Harrington K, Lacroix J, Biarent D, Joffe AR, Wensley D, Ducruet T, Hebert PC, Tucci M; TRIPICU investigators; Canadian Critical Care Trials Group; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Comparison of two red-cell transfusion strategies after pediatric cardiac surgery: a subgroup analysis. Crit Care Med. 2010 Feb;38(2):649-56. doi: 10.1097/CCM.0b013e3181bc816c. PMID 19789443
- [Background] Scrucca L, Fop M, Murphy TB, Raftery AE. mclust 5: Clustering, Classification and Density Estimation Using Gaussian Finite Mixture Models. R J. 2016 Aug;8(1):289-317. PMID 27818791